CLINICAL TRIAL: NCT07334938
Title: Effects of Far Infrared Rays and Transcutaneous Electrical Nerve Stimulation on Short Term Prognosis of Head and Neck Cancer Patients Receiving Curative Treatment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB113-052-A
Record Dates: First submitted 2025-12-16; First posted 2026-01-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Cancer (H&N)
Keywords: Head and Neck Cancer (H&N); far infrared; transcutaneous electrical nerve stimulation
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): routine care
- Transcutaneous Electrical Nerve Stimulation (TENS) (Active Comparator)
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)
- TENS Combined With Far-Infrared Therapy (Experimental)
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS); Device: Far-Infrared Therapy

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — Transcutaneous electrical nerve stimulation is applied to the neck region twice daily, in the morning and evening, for five consecutive days.
  Arms: TENS Combined With Far-Infrared Therapy; Transcutaneous Electrical Nerve Stimulation (TENS)
Device: Far-Infrared Therapy — Far-infrared therapy is applied to the neck region twice daily, in the morning and evening, for five consecutive days.
  Arms: TENS Combined With Far-Infrared Therapy

SUMMARY:
The goal of this clinical trial is to determine whether far-infrared therapy and transcutaneous electrical nerve stimulation (TENS) can improve postoperative side effects in patients with head and neck cancer. The main questions this study aims to answer are:

Can far-infrared therapy and transcutaneous electrical nerve stimulation reduce pain and improve neck range of motion?

Can far-infrared therapy and transcutaneous electrical nerve stimulation reduce inflammation?

Researchers will compare three groups:

Group A: control group; Group B: transcutaneous electrical nerve stimulation; Group C: far-infrared therapy combined with transcutaneous electrical nerve stimulation, to evaluate differences in pain, neck range of motion, and inflammation.

Participants will receive the assigned intervention in the morning and evening for five consecutive days. Outcome measurements will be conducted on the first and fifth days.

ELIGIBILITY:
Inclusion Criteria

1. Patients aged 30 to 85 years with a confirmed diagnosis of head and neck cancer.
2. Patients scheduled to undergo surgical resection.
3. Patients who are conscious, able to communicate verbally or in writing, and willing to complete questionnaires and comply with all study procedures.

Exclusion Criteria:

1. Presence of open wounds or skin lesions at the sites where transcutaneous acupoint electrical stimulation electrodes would be applied.
2. Contraindications to transcutaneous acupoint electrical stimulation, including a history of epilepsy, brain tumors, arteriovenous malformations, or implanted cardiac pacemakers or defibrillators, to avoid potential adverse effects of electrical stimulation.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Preoperative baseline (before surgery), postoperative day 10, and postoperative day 15
  Pain intensity will be assessed using a numeric rating scale (NRS), with scores ranging from 0 (no pain) to 10 (worst pain imaginable).

SECONDARY OUTCOMES:
Neck range of motion (ROM) | Preoperative baseline (before surgery), postoperative day 10, and postoperative day 15
  Active neck range of motion will be measured in degrees, including flexion, extension, bilateral rotation, and bilateral lateral flexion.
Inflammatory markers (LMR, NLR) | Preoperative baseline (before surgery), postoperative day 10, and postoperative day 15
  Inflammatory markers will be calculated from complete blood counts, including the Lymphocyte-to-monocyte ratio(LMR) and neutrophil-to-lymphocyte ratio (NLR)

CONTACTS AND LOCATIONS:
Locations (1):
- Hualien Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Hualien City, Hualien County, Taiwan

IPD SHARING:
Plan to Share IPD: No